CLINICAL TRIAL: NCT02873390
Title: A Clinical Study of PD-1 Antibody Expressing CAR-T Cells for EGFR Family Member Positive Advanced Solid Tumor
Brief Title: PD-1 Antibody Expressing CAR-T Cells for EGFR Family Member Positive Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo Cancer Hospital (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBWYKY2016-06-001/002/003
Record Dates: First submitted 2016-08-15; First posted 2016-08-19 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: PD-1 Antibody; CAR-T Cells; Advanced Malignancies
Keywords: PD-1 Antibody; CAR-T Cells; EGFR family; Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HerinCAR-PD1 cells (Experimental): Patients will receive 3 cycles of HerinCAR-PD1 cells treatment.
  Interventions: Biological: HerinCAR-PD1 cells

INTERVENTIONS:
Biological: HerinCAR-PD1 cells — herinCAR-PD1 cells transfusion: (1-5×107/kg herinCAR-PD1 + physiological saline + 0.25% human alloalbumin) 300ml for each infusion. IV (in the vein) for each infusion, 2 cycles, each cycle received one infusions on day 21, 43.

SUMMARY:
To evaluate the safety and effectiveness of cell therapy using herinCAR-PD1 cells to treat advanced cancer.

Individuals greater than or equal to 18 years of age and less than or equal to 70 years of age who have been diagnosed with relapsed or refractory cancer that has not responded to or has relapsed after standard treatment.

DETAILED DESCRIPTION:
A total of 20 patients may be enrolled over a period of 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~80 years old, male or female;
2. Life expectancy≥6 months;
3. ECOG score: 0-2;
4. Advanced Solid Tumor were diagnosed by histology and cytology;
5. Enough venous channel,no other contraindications to the separation and collection of white blood cells;
6. Immunohistochemistry and RT-PCR technology will be used to determine the positive EGFR family (including EGFR, HER2, HER4) and EGFRVIII、IGF1R protein. At least one protein expressed in immunohistochemical tumor tissue should be no less than grade 2 or 2+ scores. The levels of protein are defined as follows: (according to cell staining) : grade 0: without staining; grade 1: 1-25%; grade 2: 26-50% and grade 3: 51-100%; (According to the intensity): negative; 1+; 2+ and 3+;
7. Laboratory examination: white blood cell≥3 x 10*9/L, blood platelet count≥60 x10*9/L, hemoglobin≥85g/L; lymphocyte ≥0.7×109/L, total bilirubin less than 2.5 times of the normal level; ALT and AST less than 2.5 times of the normal level; serum creatinine less than 1.5 times of the normal level；
8. Signed informed consent；
9. Women of child-bearing age must have evidence of negative pregnancy test and be willing to practice birth control after 4 months following the cells transfusion.
10. Disease progression and the current treatment is invalid.
11. The treatment effect is not ideal after receiving 2 line therapy at least and willing to join in clinical trials

Exclusion Criteria:

1. Expected Overall survival < 6 months;
2. Patients with uncontrolled hypertension,unstable coronary disease (uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure (> Class II, NYHA), or myocardial infarction within 6 months.
3. Abnormal lung function: FEV (forced expiratory volume) < 30% prediction, DLCO (diffusing capacity of the lung for carbon monoxide) < 30% prediction, blood oxygen saturation < 90%;
4. Other serious diseases: nervous, mental disorders, immune regulatory diseases, metabolic diseases, infectious diseases, etc;
5. Unable or unwilling to provide informed consent, or fail to comply with the test requirements.
6. Uncontrolled active infection.
7. Serious chronic disease of critical organs such as kidney and liver. Kidney function more than CKD stage I,and liver function less than the Child - Pugh class B;
8. Long-term use or being used of immunosuppressive drugs with autoimmune diseases
9. Glucocorticoid is needed in a long term.
10. Currently (within 30 days) enrolled in another clinical trial.
11. Pregnancy or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
Disease control rate,(DCR) | 2 years
Overall survival | 2 years
Progress-free survival(PFS) | 2 years

SECONDARY OUTCOMES:
Quality of life | 2 years
  Questionnaire will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Jiangtao Wang, Study Director — Ningbo No.5 Hospital (Ningbo Cancer Hospital); Huajun Jin, Study Chair — Shanghai Cell Therapy Research Institute; Qijun Qian, Study Chair — Shanghai Cell Therapy Research Institute
Locations (1):
- Ningbo No.5 Hospital (Ningbo Cancer Hospital), Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No